CLINICAL TRIAL: NCT04156321
Title: Moringa Oleifera (Drumstick Leaves) for Improving Haemoglobin, Vitamin A Status and Underweight Among Adolescent Girls in Rural Bangladesh: A Quasi-experimental Study
Acronym: Moringa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-19060
Record Dates: First submitted 2019-10-17; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Assess the Impact of Moringa Leaves on Serum Heamoglobin and Vitamin A Level Among the Adolescent Girls
Keywords: Moringa, quasi-experimental, vitamin A, haemoglobin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group I (intervention) will receive 150 gm of Sajna shak/bora (Moringa) added with 25 gm concenstrated dal with 100 gm of rice as mid-morning snack in selected school 5 times a week for 6 months
  Interventions: Dietary Supplement: Moringa fry
- Control arm (No Intervention): Group II (Control) will rice, concenstrated dal and potato vaji. Both groups will receive calorie matched meal (411 kcal)

INTERVENTIONS:
Dietary Supplement: Moringa fry — School Tiffin:
  Each of the adolescent girls will receive fresh Moringa leaves (150 gram) cooked in a traditional manner as Sajna shak (stir-fried)/ bora with rice and concentrated dal once daily for 5 days during tiffin time. Sajna Stir fry and bora will be given on every alternative day. Standard questionnaire will be used to measure the compliance of food. As we are serving the food in school premises during tiffin period, it would be both unethical and socially unacceptable if few of the students from a section receive the meal. Therefore, all the students from selected section/sections will receive the daily meal. However, we will only collect information from the selected study participants who would give consent to participate in the study Each of the combination of tiffin meal will supply 411 calories in the both arm .
  Arms: Intervention

SUMMARY:
Background (brief):

1. Burden:

   Bangladesh has a population of 29.5 million adolescents, which represents nearly one-fifth of the country's total population. Adequate nutrition during this critical age period is key, and is associated with improved health and development of the future adult population, as well as that of their future off-spring bringing potential inter-generational benefits. Yet, adolescents are known to face multiple nutritional challenges related to persistent undernutrition and micronutrient deficiencies as well as rapidly rising overweight and obesity due to inadequate and inappropriate nutritional practice. A large percentage of adolescents in Bangladesh consume an inadequate diet in terms of energy content, nutrient density and diversity. To alleviate micronutrient deficiency, Moringa oleifera leaves can be used in their daily diet with a traditional manner. It contains substantial amount of protein & several essential micronutrients for growth.
2. Knowledge gap:

   Although, adolescence has been identified as a 'second window of opportunity" for correcting nutritional inadequacies and insufficient growth from childhood, however, they face multiple nutritional challenges related to persistent undernutrition and micronutrient deficiencies, particularly in resource poor countries like Bangladesh.
3. Relevance:

   About 80% of kilocalories per capita per day in Bangladesh are from micronutrient-poor foods, and 70% are from rice alone (75% for rural adolescents). A study on pregnant adolescent women showed that around 60% had low or medium dietary diversity. Among the major food groups, the routine diet of a Bangladeshi adolescent particularly lacks in protein in terms of both animal source like eggs, dairy products and plant source like legumes and nuts. Daily consumption of vitamin A-rich vegetables and fruits (other than dark-green leafy vegetables) are also inadequate. Such inadequate diet is reflected by various health outcomes. The prevalence of low Body Mass Index is 31% among married-adolescents of 15-19 years old. 13% of the adolescents are short in stature.

   Moringa leaves have a high amount of protein, and vitamins A & C, calcium, iron, potassium and zinc. It is well-known and easily cultivable in Bangladesh with limited resource. The high nutrient content of the leaves make it suitable to bring transformative changes in diet and feeding practices within the purchasing capacity of marginalized people due to its availability and affordability. Our proposed approach will assess the impact of locally available, affordable and culturally accepted Moringa leaves consumption into adolescent's regular diet to improve their nutritional status as a whole.
4. Hypothesis (if any):

   150 gm of Sajna shak /bora (Moringa) 5 days/week) will improve haemoglobin and vitamin A status of the adolescent girls after 6 months of consumption.
5. Objectives:

   The study objectives are as below:

   1.1 Primary: To assess the effect of consumption of Sajna shak/bora (Moringa) on haemoglobin and vitamin A status among the adolescent girls after 6 months of consumption 1.2 Secondary: Assess the effect of Sajna shak/bora (Moringa) on adolescent weight gain after 6 months of consumption
6. Methods:

   This will be a school-based trial. Group I (intervention) will receive 150 gm of Sajna shak/bora (Moringa) added with 25 gm concenstrated dal with 100 gm of rice as mid-morning snack in selected school 5 times a week for 6 months along with nutrition education. Group II (Control) will rice, concenstrated dal and potato vaji. Both groups will recieve calorie matched meal (411 kcal). Baseline and endline survey will be conducted. Blood sample will be collected at the baseline, at end of 3 months and at the endline. Compliance will be measured through on-spot feeding. Data on feeding, morbidity and anthropometry (height and weight) will be collected bi-monthly.
7. Outcome measures/variables:

Primary outcomes: Changes in 2 biochemical markers (haemoglobin and vitamin A).

ELIGIBILITY:
Inclusion Criteria:

-Unmarried adolescent girls aged 12-14 years will be enrolled from the selected high schools in our study,

Exclusion Criteria:

* Participants will be excluded if they are taking other nutritional supplements (vitamins and minerals) as this might affect the level of hemoglobin and other micronutrients that we intend to measure.
* Also adolescent girls with documented medical records of chronic diseases will be excluded.

Ages: 12 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 2 biochemical markers (serum haemoglobin and retinol level) | At baseline, 3 months and 6 months of intervention
  Peripheral blood samples will be collected from all participants from both intervention and control groups. Blood samples collected will be labelled with a bar-coded identification label specifically created for this study, and corresponding to study subject identification number. In this way, the laboratory could easily identify, which particular clusters are to be tested in a batch and thus minimizing the possibilities of increasing freeze/thaw cycles. A sample record/hBandover form will be filled up indicating name of the participants, ID number, sample ID number, and type of analysis to be done. The samples will be carried to the nutritional biochemistry laboratory in Dhaka in temperature controlled cooler box. Samples will be received at the laboratory and stored in a -70⁰C freezer and analyzed to estimate the blood parameters. Mean hemoglobin level (gm/dl) and serum level of retinol (mmol/l) will be measured at baseline ,3 months and after 6 months of intervention.

SECONDARY OUTCOMES:
Changes in nutritional status | At baseline, 3 months and 6 months of intervention
  Trained staff will collect anthropometric measurements (weight in kg and height in cm) monthly using established methods. Measurement would be taken at baseline, every 2 months thereafter for 6 months. Weight will be measured with minimal clothing and without any shoes and accessories in kilograms using portable Tania scale with an accuracy of accuracy of 100 g. Height will be measured at cm with height meter with 1 mm accuracy. The entire instrument will be calibrated every morning with a standard weight and height board accordingly, prior to data collection. These measurements will be standardized before and during the data collection. For our analysis of BMI status, all BMI data will be converted and categorized according to WHO cutoff points. Using the WHO BMI-for-age growth chart for girls ages 5 to 19 years, normal weight, overweight (>+1 SD, equivalent to BMI 25 kg/m obese (>+2 SD, equivalent to BMI 30 kg/m2 each study.

CONTACTS AND LOCATIONS:
Overall Officials: Mansura Khanam, Msc, Principal Investigator — Research Investigator,NCSD, icddr,b
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
icddr,b has own data sharing policy. We will follow icddr,b data sharing policy.

REFERENCES:
- See also: Related Info — https://www.icddrb.org/dmdocuments/icddrb%20Data%20Access%20Policy.pdf